CLINICAL TRIAL: NCT05749614
Title: Clinical Application of Penile Biological Vibration Threshold for Precise Use of Lidocaine Cream to Treat Primary Premature Ejaculation
Brief Title: Precise Use of Lidocaine Cream to Treat Primary Premature Ejaculation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-9941
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-03

CONDITIONS: Premature Ejaculation
Keywords: Primary premature ejaculation; Lidocaine; Arabic Index of Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Drug: Lidocaine cream
- Group 2 (Experimental)
  Interventions: Drug: Lidocaine cream

INTERVENTIONS:
Drug: Lidocaine cream — Group 1 was given 1 ml of 5% lidocaine cream on demand. They were instructed to apply the lidocaine cream evenly in a circular pattern to the glans penis without precise application to the sensitive area of the glans penis. The treatment lasted for a total of 4 weeks.
  Arms: Group 1
Drug: Lidocaine cream — Group 2 had a penile biological vibration threshold test performed to detect loci with a lower threshold. They were instructed to apply 1 ml of 5% lidocaine cream to the sensitive loci on the glans penis for 4 weeks.
  Arms: Group 2

SUMMARY:
This study aimed to evaluate the efficacy and safety of applying 5% lidocaine cream to the sensitive area of the glans penis after its precise localization under the penile biological vibration threshold test for the treatment of primary premature ejaculation.

DETAILED DESCRIPTION:
This study was a randomized, single-blind clinical controlled trial. Eighty patients diagnosed with primary premature ejaculation in an outpatient setting were included in this study. They were randomly scored into two groups. Group 1 (n = 40) was given 1 ml of 5% lidocaine cream on demand. They were instructed to apply the lidocaine cream evenly in a circular pattern to the glans penis without precise application to the sensitive area of the glans penis. The treatment lasted for a total of 4 weeks. Group 2 (n = 40) had a penile biological vibration threshold test performed to detect loci with a lower threshold. They were instructed to apply 1 ml of 5% lidocaine cream to the sensitive loci on the glans penis for 4 weeks. Lidocaine cream was applied topically or uniformly to the glans penis 20 minutes before planned intercourse in both groups and washed off 10 minutes after application. Using intravaginal ejaculation before and after treatment latency, the Arabic Index of Premature Ejaculation, Premature Ejaculation Diagnostic Tool, and the International Index of Erectile Function Scale scores were combined to assess the efficacy and side effects before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* adult male (19-60 years old); stable partner for ≥3 months; Premature Ejaculation Diagnostic Tool (PEDT) score ≥ 11; penile biological vibration threshold test suggesting the presence of sensitive sites on the glans penis (vibration threshold < 30 levels); no history of long-term use of specific medications; normal sex hormone levels; and no genital or secondary ejaculation. There was no history of long-term use of specific drugs, normal sex hormone levels, and genital or secondary sexual characteristics abnormalities.

Exclusion Criteria:

* (1) those with abnormal or malformed genital development; (2) those with allergic reactions to local anesthetics; (3) those who had been treated with central nervous system drugs or PE in the last 3 months; (4) those with a history of long-term alcohol abuse and trauma such as neurological and pelvic fractures; (5) those with long-term use of hypotensive drugs, diuretics, and sedative drugs (6) patients with a history of previous surgery and trauma to the reproductive system; (7) patients with PE due to hypogonadism, thyroid disease, and abnormal lipid metabolism.

Ages: 19 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Arabic Index of Premature Ejaculation (AIPE) | through study completion,an average of 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Luopei Wei, Hangzhou, Zhejiang, China